CLINICAL TRIAL: NCT04672031
Title: Tight Versus Standard Glycemic Targets for Pregnant Women With Gestational Diabetes and Type 2 Diabetes
Brief Title: Glycemic Targets for Pregnant Women With GDM and T2DM
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Southern California (Other)
Responsible Party: Principal Investigator, Brendan Grubbs, Assistant Professor, University of Southern California
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: APP-20-06210
Record Dates: First submitted 2020-12-08; First posted 2020-12-17 (Actual); Last update posted 2023-05-11 (Actual); Status verified 2023-05

CONDITIONS: Diabetes Mellitus in Pregnancy; Diabetes, Gestational; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes, Gestational; Diabetes Mellitus, Type 2

STUDY DESIGN:
Intervention Model Description: Eligible women will be randomized at a 1:1 ratio (using block randomization) into either the control arm or the intervention arm. It is understood that study participants, physicians, and nurse-educators cannot be blinded to group allocation. The randomization process will proceed as follows. A primary randomization model assigning patients to the "New Target" versus the "Standard Target" will be created for the one center (LAC+USC), and permuted-block randomization with random allocation will be used. The investigators will be blinded to the block size. The generation of randomization codes will be performed using SAS statistical software, v. 9.3, Cary, NC. A validation test will be performed to assure that treatment balance is achieved within the entire study.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Arm (No Intervention): Patients in the control arm will be instructed to check blood sugars seven times per day: fasting, pre-prandial, and 1 hour after each meal. The glycemic targets for the control arm will be defined as follows: fasting ≤95 mg/dL, pre-prandial ≤95 mg/dL, and 1-hour postprandial ≤140 mg/dL (i.e. conventional targets). Patients who do not achieve glycemic goals with diet and exercise will be started on medical therapy (metformin or insulin) at the discretion of a maternal-fetal medicine subspecialist and endocrinologist.
- Interventional Arm (Experimental): Patients in the experimental arm will be instructed to check blood sugars seven times per day: fasting, pre-prandial, and 1 hour after each meal. The glycemic targets for the intervention arm will be defined as follows: fasting ≤80 mg/dL, pre-prandial ≤80 mg/dL, and 1-hour postprandial ≤110 mg/dL. Patients who do not achieve glycemic goals with diet and exercise will be started on medical therapy (metformin or insulin) at the discretion of a maternal-fetal medicine subspecialist and endocrinologist.
  Interventions: Other: Glycemic Targets

INTERVENTIONS:
Other: Glycemic Targets — The intervention is glycemic targets that are lower than those currently recommended by ADA and ACOG: fasting ≤80 mg/dL, pre-prandial ≤80 mg/dL, and 1-hour postprandial ≤110 mg/dL instead of fasting ≤95 mg/dL, pre-prandial ≤95 mg/dL, and 1-hour postprandial ≤140 mg/dL.
  Arms: Interventional Arm

SUMMARY:
The purpose of this randomized clinical trial is to determine whether glycemic targets that are lower than those currently recommended by the American Diabetes Association (ADA) and the American College of Obstetricians and Gynecologists (ACOG) would improve overall outcomes in pregnant patients with diabetes. Eligible pregnant women with a diagnosis of gestational diabetes or Type 2 diabetes will be randomized into either routine care with glycemic targets as currently recommended by ADA and ACOG (control arm), or more aggressive care with lower glycemic targets that more closely resemble normoglycemia in pregnancy (intervention arm). The glycemic targets for the control arm will be defined as follows: fasting ≤95 mg/dL, pre-prandial ≤95 mg/dL, and 1-hour postprandial ≤140 mg/dL. The glycemic targets for the intervention arm will be defined as follows: fasting ≤80 mg/dL, pre-prandial ≤80 mg/dL, and 1-hour postprandial ≤110 mg/dL. The primary outcome will be a 250-gram difference in birth weight between the two study arms. Secondary maternal and neonatal outcomes of interest will also be compared between the two study arms.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women with a singleton gestation
* 18 years or older
* Diagnosis of gestational diabetes (prior to 34 weeks gestational age) or Type 2 diabetes

Exclusion Criteria:

* Diagnosed with gestational diabetes at or beyond 34 weeks gestational age
* Type 1 diabetes
* Diabetic retinopathy
* Diabetic nephropathy
* Diabetic vasculopathy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2021-07-08 (Actual); Primary Completion 2023-07 (Estimated); Study Completion 2023-07 (Estimated)

PRIMARY OUTCOMES:
Difference in birth weight | 41 weeks gestation
  250-gram difference in birth weight

SECONDARY OUTCOMES:
Total prenatal care visits | 41 weeks gestation
  Total number of prenatal care visits during pregnancy
Prenatal care visits after enrollment | 41 weeks gestation
  Number of prenatal care visits after enrollment
Prenatal care visits: log/glucometer | 41 weeks gestation
  Number of prenatal care visits with log/glucometer available for RN or MD to review
Prenatal care visits: targets met | 41 weeks gestation
  Number of prenatal care visits in which patient met blood sugar targets
Prenatal care visits: intervention | 41 weeks gestation
  Number of prenatal care visits in which an intervention for blood sugars was recommended (e.g. starting medication or changing medication dose)
Symptomatic hypoglycemia | 41 weeks gestation
  Frequency of symptomatic hypoglycemia episodes (hypoglycemia defined as <70 mg/dL per ADA)
Asymptomatic hypoglycemia | 41 weeks gestation
  Frequency of asymptomatic hypoglycemia episodes (hypoglycemia defined as <70 mg/dL per ADA)
A1c enrollment | At time of enrollment (up to 34 weeks gestation)
  Hemoglobin A1c at the time of enrollment
A1c 36 weeks | At 36 weeks gestational age
  Hemoglobin A1c at 36 weeks gestational age
Lowest recorded blood sugar | 41 weeks gestation
  Lowest recorded blood sugar during prenatal care
Highest recorded blood sugar | 41 weeks gestation
  Highest recorded blood sugar during prenatal care
Average recorded blood sugar | 41 weeks gestation
  Average recorded blood sugar during prenatal care
Weekly compliance | 41 weeks gestation
  Average number of blood sugar checks actually performed each week
Weekly target assessment | 41 weeks gestation
  % of blood sugars within goal each week
Diabetes medication | 41 weeks gestation
  Did the patient need diabetes medication (including oral agents and insulin) during antepartum period?
Intrapartum insulin | From onset of induction/labor until delivery
  Did the patient need insulin during the intrapartum period?
Gestational weight gain | 41 weeks gestation
  Total weight gain during pregnancy in kilograms
Antepartum admission | 41 weeks gestation
  Was the patient ever admitted to antepartum service for any indication, including poorly-controlled diabetes or diabetes-related complication?
Corticosteroids | 41 weeks gestation
  Did the patient receive antenatal corticosteroid treatment?
Oligohydramnios | 41 weeks gestation
  Amniotic fluid index <5 cm or maximum vertical pocket <2cm
Polyhydramnios | 41 weeks gestation
  Amniotic fluid index >24cm or maximum vertical pocket >8cm
Fetal growth restriction | 41 weeks gestation
  Ultrasonographic estimated fetal weight or abdominal circumference <10% for gestational ag
Gestational age at delivery | During intrapartum admission to Labor & Delivery
  Gestational age at delivery
Induction of labor | During intrapartum admission to Labor & Delivery
  Did the patient undergo induction of labor?
Mode of delivery | During intrapartum admission to Labor & Delivery
  primary cesarean section, repeat cesarean section, vaginal delivery, vaginal delivery with vacuum, vaginal delivery with forceps
Cesarean indication | During intrapartum admission to Labor & Delivery
  If the patient had cesarean delivery, what was the indication?
TOLAC | During intrapartum admission to Labor & Delivery
  Did the patient attempt a trial of labor after cesarean?
Blood loss | During intrapartum admission to Labor & Delivery
  Quantitative blood loss (or estimated if quantitative is unknown) in cc's
3rd or 4th degree laceration | During intrapartum admission to Labor & Delivery
  3rd or 4th degree perineal laceration
PIH | From 20 weeks gestation until 30 days postpartum
  Pregnancy-induced hypertension (gestational hypertension, preeclampsia, HELLP syndrome)
Hypertensive emergency | From conception until 30 days postpartum
  Did the patient have severe-range blood pressures require antihypertensive medication?
Chorioamnionitis | During intrapartum admission to Labor & Delivery
  Chorioamnionitis
Endometritis | Within 30 days postpartum
  Endometritis
VTE | From conception until 30 days postpartum
  Venous thromboembolism: deep venous thrombosis or pulmonary embolism
Length of stay (maternal) | From admission to Labor & Delivery until discharge from postpartum
  Length of hospital admission for labor, delivery, and postpartum
Postpartum readmission | Within 30 days postpartum
  Did the patient get readmitted within 30 days of delivery?
Postpartum wound complication | Within 30 days postpartum
  Cesarean wound infection of dehiscence, perineal laceration breakdown
Cardiac complications | From conception until 30 days postpartum
  Did the patient develop any cardiac complications such as arrhythmias or cardiomyopathy?
Seizures | From conception until 30 days postpartum
  Did any maternal seizures occur during the pregnancy or postpartum?
Macrosomia | Within 24 hours of birth
  Birth weight >4000 grams
LGA | Within 24 hours of birth
  Large for gestational age (birth weight ≥90% for gestational age)
SGA | Within 24 hours of birth
  Small for gestational age (birth weight <10% for gestational age)
Shoulder dystocia | During intrapartum admission to Labor & Delivery
  Shoulder dystocia
Apgar | 5 minutes after birth
  5-minute Apgar score
Cord gas pH <7.0 | Within 24 hours of birth
  Did the baby have a cord blood gas pH <7.0?
Base excess | Within 24 hours of birth
  What was the base excess on the cord blood gas?
Neonatal blood glucose | Within 24 hours of birth
  What was the neonatal serum blood glucose at birth?
RDS | Within 30 days of delivery
  Neonatal respiratory distress syndrome
TTN | Within 30 days of delivery
  Transient tachypnea of the newborn
Hyperbilirubinemia | Within 30 days of delivery
  Neonatal hyperbilirubinemia (as defined in AAP 2004 Clinical Practice Guideline "Management of Hyperbilirubinemia in the Newborn Infant 35 or More Weeks of Gestation")
Neonatal sepsis | Within 30 days of delivery
  Neonatal sepsis
NICU | Within 30 days of delivery
  NICU admission
Length of stay (neonatal) | From birth until discharge (up to 1 year)
  How many days after birth did the neonate stay in the hospital?
Congenital anomaly | Within 30 days of delivery
  Congenital anomaly
IUFD or stillbirth | From conception until delivery
  Intrauterine fetal demise or stillbirth

CONTACTS AND LOCATIONS:
Locations (1):
- Los Angeles County + University of Southern California Medical Center (LAC+USC), Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Macrosomia: ACOG Practice Bulletin, Number 216. Obstet Gynecol. 2020 Jan;135(1):e18-e35. doi: 10.1097/AOG.0000000000003606. PMID 31856124
- [Background] ACOG Practice Bulletin No. 190: Gestational Diabetes Mellitus. Obstet Gynecol. 2018 Feb;131(2):e49-e64. doi: 10.1097/AOG.0000000000002501. PMID 29370047
- [Background] ACOG Practice Bulletin No. 190 Summary: Gestational Diabetes Mellitus. Obstet Gynecol. 2018 Feb;131(2):406-408. doi: 10.1097/AOG.0000000000002498. PMID 29370044
- [Background] Metzger BE, Coustan DR. Summary and recommendations of the Fourth International Workshop-Conference on Gestational Diabetes Mellitus. The Organizing Committee. Diabetes Care. 1998 Aug;21 Suppl 2:B161-7. No abstract available. PMID 9704245
- [Background] Hernandez TL. Glycemic targets in pregnancies affected by diabetes: historical perspective and future directions. Curr Diab Rep. 2015 Jan;15(1):565. doi: 10.1007/s11892-014-0565-2. PMID 25398204
- [Background] Fraser R. Diabetic control in pregnancy and intrauterine growth of the fetus. Br J Obstet Gynaecol. 1995 Apr;102(4):275-7. doi: 10.1111/j.1471-0528.1995.tb09130.x. No abstract available. PMID 7612507
- [Background] Dandona P, Besterman HS, Freedman DB, Boag F, Taylor AM, Beckett AG. Macrosomia despite well-controlled diabetic pregnancy. Lancet. 1984 Mar 31;1(8379):737. doi: 10.1016/s0140-6736(84)92248-7. No abstract available. PMID 6143065
- [Background] Combs CA, Gunderson E, Kitzmiller JL, Gavin LA, Main EK. Relationship of fetal macrosomia to maternal postprandial glucose control during pregnancy. Diabetes Care. 1992 Oct;15(10):1251-7. doi: 10.2337/diacare.15.10.1251. PMID 1425084
- [Background] Hernandez TL, Friedman JE, Van Pelt RE, Barbour LA. Patterns of glycemia in normal pregnancy: should the current therapeutic targets be challenged? Diabetes Care. 2011 Jul;34(7):1660-8. doi: 10.2337/dc11-0241. No abstract available. PMID 21709299
- [Background] Thompson DM, Dansereau J, Creed M, Ridell L. Tight glucose control results in normal perinatal outcome in 150 patients with gestational diabetes. Obstet Gynecol. 1994 Mar;83(3):362-6. PMID 8127526
- [Background] Carpenter MW, Coustan DR. Criteria for screening tests for gestational diabetes. Am J Obstet Gynecol. 1982 Dec 1;144(7):768-73. doi: 10.1016/0002-9378(82)90349-0. PMID 7148898
- [Background] Buchanan TA, Kjos SL, Montoro MN, Wu PY, Madrilejo NG, Gonzalez M, Nunez V, Pantoja PM, Xiang A. Use of fetal ultrasound to select metabolic therapy for pregnancies complicated by mild gestational diabetes. Diabetes Care. 1994 Apr;17(4):275-83. doi: 10.2337/diacare.17.4.275. PMID 8026282
- [Background] Kjos SL, Schaefer-Graf U, Sardesi S, Peters RK, Buley A, Xiang AH, Bryne JD, Sutherland C, Montoro MN, Buchanan TA. A randomized controlled trial using glycemic plus fetal ultrasound parameters versus glycemic parameters to determine insulin therapy in gestational diabetes with fasting hyperglycemia. Diabetes Care. 2001 Nov;24(11):1904-10. doi: 10.2337/diacare.24.11.1904. PMID 11679455
- [Background] American Diabetes Association. 14. Management of Diabetes in Pregnancy: Standards of Medical Care in Diabetes-2020. Diabetes Care. 2020 Jan;43(Suppl 1):S183-S192. doi: 10.2337/dc20-S014. PMID 31862757
- [Result] American Academy of Pediatrics Subcommittee on Hyperbilirubinemia. Management of hyperbilirubinemia in the newborn infant 35 or more weeks of gestation. Pediatrics. 2004 Jul;114(1):297-316. doi: 10.1542/peds.114.1.297. PMID 15231951
- [Result] American Diabetes Association. 6. Glycemic Targets: Standards of Medical Care in Diabetes-2019. Diabetes Care. 2019 Jan;42(Suppl 1):S61-S70. doi: 10.2337/dc19-S006. PMID 30559232